CLINICAL TRIAL: NCT02039687
Title: A Double Blind, Placebo Controlled Phase 2 Dose Ranging Study of the Effects of ARA 290 on Corneal Nerve Fiber Density and Neuropathic Symptoms of Subjects With Sarcoidosis
Brief Title: Study of Efficacy of ARA 290 on Corneal Nerve Fiber Density and Neuropathic Symptoms of Subjects With Sarcoidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Araim Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APCP-112
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Neuropathy of Sarcoidosis
Keywords: neuropathy; sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — cibinetide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 mg per day ARA 290 (Experimental): 1 mg ARA 290 administered subcutaneously for 28 consecutive days
  Interventions: Drug: ARA 290
- 4 mg per day ARA 290 (Experimental): 4 mg ARA 290 administered subcutaneously for 28 consecutive days
  Interventions: Drug: ARA 290
- 8 mg per day ARA 290 (Experimental): 8 mg ARA 290 administered subcutaneously for 28 consecutive days
  Interventions: Drug: ARA 290
- placebo (Placebo Comparator): 1 mL placebo administered subcutaneously for 28 consecutive days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ARA 290 — A small peptide that activates the innate repair receptor to induce anti-inflammatory and tissue repair mechanisms.
  Other Names: pHSBP, Cibinetide
  Arms: 1 mg per day ARA 290; 4 mg per day ARA 290; 8 mg per day ARA 290
Other: Placebo — Formulation buffer
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether ARA 290, a new class of compound, is effective in the treatment of the neuropathic symptoms of sarcoidosis. Brief interaction of ARA 290 with the innate repair receptor results in anti-apoptotic and anti-inflammatory activities in myriad of cells, tissues and organs throughout the body to activate repair mechanisms and accelerate healing, including the nerve damage that can be associated with sarcoidosis. In this study, subjects with sarcoidosis and symptoms of small fiber neuropathy will administered ARA 290 or placebo by subcutaneous injection daily for 28 days. In addition to monitoring the safety of the treatment, the symptoms of the subjects will be assessed with several questionnaires, function tests, and measurement of nerve fibers in their cornea and skin (via a non-invasive test and a biopsy, respectively). The total participation time for each patient will be 16 weeks.

DETAILED DESCRIPTION:
This was a double-blind, randomized, placebo-controlled study to assess the effects of daily SC administration of ARA 290 at a dose of 1 mg, 4 mg, or 8 mg or placebo on corneal nerve fiber density of subjects with sarcoidosis and neuropathic symptoms consistent with small fiber neuropathy. The safety of these doses was also assessed.

Up to 64 subjects with sarcoidosis and symptoms of small fiber neuropathy were planned to be enrolled in the study. Subjects determined to be eligible at the screening visit were asked to return to the study site for the start of the treatment period (Visit 1, study day 1) within 28 days of screening. Subjects who were not able to return for Visit 1 within 28 days of the screening visit could be rescreened. At Visit 1, the subjects were randomized to one of 4 treatment groups (approximately 16 subjects per group): 1 mg, 4 mg, or 8 mg of ARA 290 or placebo. The study drug (ARA 290 or placebo) was to be administered daily for 28 days via SC injection. The first injection of study drug was administered at the study site at Visit 1. After the first injection, the subjects were required to stay at the research site for 1 hour post dose for safety observation and recording of any adverse events (AEs). The subjects were trained for self-injection of the study drug and asked to self-administer the study medication daily at home before breakfast for the remaining treatment period using the supplied individual vials and disposable insulin needles and syringes.

The subjects were asked to visit the study site after 14 ± 2 days of dosing (Visit 2) and at the end of the treatment period Day 28 ± 2 (Visit 3). Additionally, the study personnel contacted the subjects by telephone at study days 7 and 21. Following the treatment period the subjects were followed-up for a further 12 weeks (until study day 112). During this period the subjects visited the study site at Day 56 ± 2 days (Visit 4) and study personnel contacted the subjects by telephone at study days 35 and 42 and biweekly from study days 70 to 112. The duration of study participation for each subject was 16 weeks. Throughout the study the subjects were asked to complete several questionnaires regarding general health and well-being, pain, fatigue and neuropathic symptoms. Further assessments included the 6MWT, and determination of nerve fiber density. If feasible at the site, quantitative sensory and cardiac autonomic reflex testing were to be performed.

The protocol was later amended to administer the Columbia-Suicide Severity Rating Scale (C-SSRS). Any positive results for active suicidal ideation and behavior, based on evaluation of the C-SSRS questionnaire, were reported as AEs. During the treatment period the subjects were also asked to complete a diary card to document compliance. Safety assessments included the documentation of AEs, vital signs and electrocardiogram (ECG), safety laboratory, physical examination and a test for ARA 290 antibodies.

ELIGIBILITY:
Inclusion Criteria:

• Established diagnosis of sarcoidosis with both of the following two criteria:

1. Score of 4 or greater on Brief Pain Inventory "pain now" or "average pain" questions (BPI; 0 (least discomfort)-10 (worst discomfort))
2. Discomfort defined as distal pain/discomfort plus one of the following: 1) dysesthesia, 2) burning/painful feet worsening at night, or 3) intolerance of sheets or clothes touching the legs or feet

AND either of the following two criteria

1. Corneal nerve fiber density reduced compared to normal (i.e., greater than 1 standard deviation less than the mean of a normative population)
2. A previous skin biopsy (obtained within the prior 2 years) showing a reduced intraepidermal nerve fiber density ((i.e., greater than 1 standard deviation less than the mean of a normal age and gender relevant population)

In addition, subjects must:

* Be able to read and understand the written consent form, complete study-related procedures, and communicate with the study staff
* Be willing to comply with study restrictions
* Be willing to check in with the study center via the telephone
* Between 18 and 70 years of age (inclusive)
* Body Mass Index (BMI) < 40 kg/m2 (inclusive)
* If female of childbearing potential, a negative urine pregnancy test at screening and acceptable contraception will be maintained during the screening and dosing period and 1 month beyond. Acceptable contraception consists of hormonal methods such as oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full cycle (based on the subject's usual menstrual cycle period) before study entry, intrauterine device (IUD), or double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream).
* Able to complete self-administered questionnaires (RAND-36, SFNSL, BPI, FAS, NPSI)
* Refrigerator and freezer at home for storage of study medication.

Exclusion Criteria:

* Clinically relevant abnormal history of physical and mental health other than conditions related to sarcoidosis, as determined by medical history taking (as judged by the investigator)
* Clinically relevant abnormal laboratory results, vital signs, or physical findings other than conditions related to sarcoidosis or could interfere with conduct of 6-minute walk assessment (as judged by the investigator)
* Other medical conditions known to be associated with small nerve fiber loss, except for diabetes in good control (as judged by the investigator)
* Known clinically relevant abnormalities in ECG (as judged by the investigator)
* Illicit drug abuse or excessive alcohol consumption (as judged by the investigator)
* History of serious malignancy within the last 5 years other than a basal cell or squamous cell carcinoma of the skin that has been removed
* History of severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food (as judged by the investigator)
* Anti-TNF therapy, other biological anti-inflammatory agents, or immunoglobulins administered within the 3 months prior to screening.
* Use of erythropoiesis stimulating agents within the two months prior to screening or during the trial
* Participation in an investigational drug trial in the 3 months prior to administration of the initial dose of study drug or more than 4 times in the calendar year preceding study enrollment
* Inadequate venous accessibility as judged by clinicians (physician or nurse)
* Inability or unwillingness to self-administer ARA 290 via subcutaneous injections (or not have access to home health care for assistance in administration)
* If female, pregnant or breast-feeding
* Any other condition that in the opinion of the investigator would complicate or compromise the study, or the well-being of the subject

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Brines, MD, PhD, Study Director — Araim Pharmaceuticals, Inc.
Locations (2):
- Cleveland Clinic, Cleveland, Ohio, United States
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 mg Per Day ARA 290 | 4 mg Per Day ARA 290 | 8 mg Per Day ARA 290 | Placebo
Started | 16 | 16 | 16 | 16
Completed | 16 | 15 | 13 | 16
Not Completed | 0 | 1 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — treatment assignment could not be confir | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg Per Day ARA 290 | 4 mg Per Day ARA 290 | 8 mg Per Day ARA 290 | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 14 | 16 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (7.47) | 51.8 (10.75) | 52.2 (9.17) | 47.8 (10.66) | 50.8 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 6 | 9 | 32
  Male | 8 | 7 | 8 | 7 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 16 | 15 | 14 | 16 | 61
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Corneal Nerve Fiber Area
Description: Measurement of corneal nerve fiber area is a non-invasive procedure performed at baseline and at the end of dosing and at 12 weeks follow-up. The nerve fiber area in sarcoidosis patients is reduced compared to normal humans, a measurement of small fiber loss.
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: µm^2
Arm/Group | 1 mg Per Day ARA 290 | 4 mg Per Day ARA 290 | 8 mg Per Day ARA 290 | Placebo
Number analyzed (Participants) | 16 | 16 | 14 | 16
µm^2 | -64.3 (759.9) | 533.8 (1110.02) | 203.8 (641.2) | -170.0 (633.0)

2. Secondary Outcome: Change in the 6 Minute Walk Test
Description: Measurement of the distance a patient can walk in 6 minutes
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | 1 mg Per Day ARA 290 | 4 mg Per Day ARA 290 | 8 mg Per Day ARA 290 | Placebo
Number analyzed (Participants) | 16 | 16 | 14 | 16
meters | 19.3 (79.27) | 17.7 (40.29) | 18.2 (47.9) | 1.2 (38.56)

3. Secondary Outcome: Change in Intra-epidermal Nerve Fiber Density (IENFD)
Description: Measurement of small fiber density in skin biopsies. Density is reduced in sarcoidosis patients, an indication of neuropathy.
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: fibers/mm
Arm/Group | 1 mg Per Day ARA 290 | 4 mg Per Day ARA 290 | 8 mg Per Day ARA 290 | Placebo
Number analyzed (Participants) | 16 | 16 | 14 | 16
fibers/mm | 0.5 (1.58) | 0.4 (2.28) | -0.3 (1.81) | 0.8 (1.13)

4. Secondary Outcome: Change in the Scores of the SFNSL, BPI, NPSI, and FAS Questionnaires
Description: Change in mean score from baseline to Day 28 is recorded for each outcome. Brief Pain Inventory (BPI), Pain Severity - scale of 0 (no pain) to 10 (worst pain imaginable) in 4 time frames, averaged.
  BPI, Pain Interference - scale of 0 (does not interfere) to 10 (completely interferes) how pain interferes with 7 lifestyle parameters, averaged.
  Small Fiber Neuropathy Screening List (SFNSL) - scale of 0 to 84 (higher score indicates greater neuropathy), sum of 21 questions.
  Neuropathic Pain Symptom Inventory (NPSI) - scale of 0 (least pain) to 10 (most pain) in 10 questions, summed. Total score range from 0 to 100.
  Fatigue Assessment Scale (FAS) - scale of 1 (never) to 5 (always) in 10 questions related to fatigue, summed. Total score range from 0 to 50, with 0 being the best possible score and 50 the worst..
Time Frame: Baseline to 28 days
Population: Questionnaires incomplete for some subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg Per Day ARA 290 | 4 mg Per Day ARA 290 | 8 mg Per Day ARA 290 | Placebo
Number analyzed (Participants) | 16 | 16 | 14 | 16
units on a scale
  BPI - Pain Severity: number analyzed (Participants) | 16 | 15 | 13 | 16
  BPI - Pain Severity | -0.594 (1.6680) | -1.167 (1.6894) | -1.115 (1.7067) | -0.922 (1.4429)
  BPI - Pain Interference: number analyzed (Participants) | 16 | 15 | 13 | 16
  BPI - Pain Interference | -1.187 (1.9453) | -1.657 (1.6482) | -1.308 (2.4403) | -1.732 (2.2174)
  SFNSL: number analyzed (Participants) | 16 | 15 | 13 | 15
  SFNSL | -4.9 (8.87) | -8.7 (14.17) | -5.5 (7.09) | -7.3 (9.50)
  NPSI: number analyzed (Participants) | 16 | 14 | 13 | 16
  NPSI | -12.31 (16.074) | -14.50 (17.887) | -8.38 (12.699) | -12.88 (13.803)
  FAS: number analyzed (Participants) | 16 | 15 | 13 | 16
  FAS | -2.6 (5.52) | -2.1 (5.38) | -3.1 (5.27) | -2.2 (6.00)

5. Secondary Outcome: Frequency of Adverse Events, Serious Adverse Events, and Laboratory Parameters
Description: Patients reporting at least one treatment emergent adverse event (TEAE) or serious TEAE
Time Frame: Continuous reporting from baseline through 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg Per Day ARA 290 | 4 mg Per Day ARA 290 | 8 mg Per Day ARA 290 | Placebo
Number analyzed (Participants) | 16 | 16 | 14 | 16
Participants
  Patients reporting at least one TEAE | 14 | 11 | 12 | 12
  Patients reporting at least one serious TEAE | 2 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 28 day treatment with 84 day follow up
Arm/Group | 1 mg Per Day ARA 290 | 4 mg Per Day ARA 290 | 8 mg Per Day ARA 290 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/16 | 0/16 | 1/14 | 0/16
Other Adverse Events (participants affected / at risk) | 14/16 | 11/16 | 12/14 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg Per Day ARA 290 (N=16) | 4 mg Per Day ARA 290 (N=16) | 8 mg Per Day ARA 290 (N=14) | Placebo (N=16)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Tightness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small Bowel Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg Per Day ARA 290 (N=16) | 4 mg Per Day ARA 290 (N=16) | 8 mg Per Day ARA 290 (N=14) | Placebo (N=16)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness exertional (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retrograde Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (4) | 2 (2) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tearfulness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Accommodation disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sticky skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less